CLINICAL TRIAL: NCT04643496
Title: Post-operative CRP Monitoring After Ileo-colic Resection in Crohn's Disease Patients
Brief Title: CRP Monitoring After ICR in CD Patients
Acronym: C-ICR-CD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0632
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2020-11

CONDITIONS: Crohn Disease; Ileocolic Resection
Keywords: Laparoscopy; C-reactive protein; Postoperative outcomes; Intra-abdominal septic complications
MeSH Terms: conditions — Crohn Disease | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients requiring ileocolic resection for Crohn disease.: All consecutive patients requiring an ileocolic resection for Crohn disease, between January 2010 and March 2020 at the Digestive Surgery Units of CHU Montpellier.
  Interventions: Procedure: Laparoscopic or open Ileocolic resection

INTERVENTIONS:
Procedure: Laparoscopic or open Ileocolic resection — Laparoscopic or open Ileocolic resection

SUMMARY:
Aim: The aim of this study was to assess the accuracy of the C-reactive protein as an early predictor of intra-abdominal septic complicationss after ileocolic resection for Crohn disease.

Methods: Data collected between January 2010 and March 2020 will be analyzed. Informations about preoperative, peroperative and post operative will be collected. The outcome after surgery will be analysed according to the comprehensive complication index.

DETAILED DESCRIPTION:
In colorectal surgery, inflammatory markers (CRP, PCT) are used systematically in the postoperative period as an early predictor of postoperative complications and in particular the prediction of anastomotic leaks and intra-abdominal septic complications.

Indeed, the occurrence of an anastomotic leak (5 to 15% of cases) involves the introduction of antibiotics, the carrying out of invasive procedures which can go as far as reoperation (and the establishment of ostomy) and always increases the length of stay and the cost of hospitalization. It is therefore essential to benefit from the most sensitive and specific tools to detect this serious and sometimes lethal complication at an early stage.

Numerous studies have evaluated and demonstrated the value of monitoring the CRP in the early postoperative period to detect the occurrence of an anastomotic leak. However, the majority of these studies presented heterogeneous populations for two reasons: all types of colorectal surgery interventions were included (right colectomy, transverse colectomy, left colectomy and anterior resection of the rectum) and multiple surgical indications were taken into account (colorectal cancer, inflammatory bowel disease, colonic diverticulosis).

In addition, a 2015 study comparing the postoperative monitoring of markers of inflammation after ileocolic resection of patients with, on the one hand, Crohn's disease and, on the other, colon cancer showed a greater inflammatory reaction in patients with Crohn's disease (in particular on POD1, 4, 5 and 6) without identifying a threshold value. This increased inflammatory response can be explained by a greater inflammatory state than in the general population: bacterial translocation due to an alteration of the mucosal barrier aggravated by immunodeficiency.

It thus appears that the cut-off values usually used (170-175 mg/l on POD3 and 125mg/l on POD4) are probably not suitable for the postoperative monitoring of these patients and for prediction of intra-abdominal septic complications.

No study to date has identified a threshold value of postoperative CRP that can predict the occurrence of postoperative anastomotic fistula and intra-abdominal septic complications after ileocecal resection for Crohn's disease.

ELIGIBILITY:
Inclusion criteria:

* Patients who underwent an ileocolic resection for Crohn disease
* Patient ≥18 years old

Exclusion Criteria:

- Patient who reject the study protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective review of collected data including all consecutive patients requiring an ileocolic resection for Crohn disease between January 2010 and March 2020 at the Digestive Surgery Units of CHU Montpellier.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of intra-abdominal septic complications | 90 days (after surgery)
  Rate of intra-abdominal septic complications

SECONDARY OUTCOMES:
Anastomotic leak rate | 90 days (after surgery)
  Anastomotic leak rate
Rate ofMorb idity according to the Clavien Dindo Classification | 90 days (after surgery)
  Morbidity according to the Clavien Dindo Classification
Rate of Mortality | 90 days (after surgery)
  Mortality
Number of Participants with Hemorragic complications | 90 days (after surgery)
  Hemorragic complications
Reoperation rate | 90 days (after surgery)
  Reoperation rate
Post-operative rate of stomy | 90 days (after surgery)
  Post-operative rate of stomy
Readmission rate | 90 days (after surgery)
  Readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC